CLINICAL TRIAL: NCT03403062
Title: Prognostic Value of Red Cell Distribution Width (RDW) in Neonatal Sepsis in Patients Admitted at Assiut University Children Hospital.
Brief Title: Prognostic Value of Red Cell Distribution Width (RDW) in Neonatal Sepsis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, mariam nagy gamil, Principal investigator, Assiut University
Other Study IDs: RDW and neonatal sepsis
Record Dates: First submitted 2017-12-13; First posted 2018-01-18 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Neonatal SEPSIS
Keywords: Sepsis; red cell distribution width (RDW); Late onset sepsis (LOS); Early onset sepsis (EOS)
MeSH Terms: conditions — Neonatal Sepsis; Sepsis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. Evaluate the relationship of RDW and severity and mortality in patients with neonatal sepsis .
2. Using RDW as a simple, inexpensive, applicable and rapid test to detect prognosis of neonatal sepsis .

DETAILED DESCRIPTION:
Sepsis is defined as a life-threatening condition caused by a dysregulated host response to infection. Sepsis is responsible for approximately 45% of neonatal emergencies and is a leading cause of neonatal mortality and morbidity, accounting for 14% of deaths in that age group.

The early symptoms and signs of neonatal sepsis are usually mild and nonspecific but can rapidly progress to septic shock, disseminated intravascular coagulation(DIC), and death. It is therefore of paramount importance to find a tool for prediction of infants who are more likely to experience a worse clinical outcome so that closer monitoring and more aggressive treatment would be offered to them.

Early-onset sepsis (EOS) is usually due to transplacental, ascending, or intrapartum transmission in the perinatal period shortly before or during birth, up to postnatal (PN) 7 days. Late-onset sepsis (LOS) is acquired by horizontal transmission in the home, hospital, or in the community after PN day.

Timely diagnosis and prompt institution of antimicrobial therapy are essential in order to mitigate the high case fatality and to avert morbidity associated with late-onset neonatal sepsis. In the latest years, biochemical markers are important in research areas in neonatal infections. Inflammatory cascade as response to an infection comprise many elevated markers, frequently used for diagnosis and monitoring of sepsis.

Numerous molecules have been studied as potentially useful prognostic markers in neonatal sepsis. These include C-reactive protein (CRP), procalcitonin, IL-6, IL-8, CD64, and soluble E- selectin.

The red cell distribution width (RDW) is a marker, which has been studied in neonatal sepsis. The RDW is a measure of variability of red blood cells in size (anisocytosis) and is routinely evaluated as a part of complete blood count. The RDW may be elevated in conditions of ineffective production, or increased destruction of red blood cells, which commonly occur in inflammatory or infectious situations.

Red cell distribution width has been classically used as a screening index for iron deficiency anemia. However, a growing body of evidence indicates that this simple marker can have a role in predicting adverse outcome in sepsis as well as in diverse clinical situations, including coronary artery disease, heart failure,acute pancreatitis, malignancy, infective endocarditis, peritoneal dialysis, and in critically ill children in general.

The pathophysiology of the elevation of RDW in these patients is not well known, but it has been reported that elevated RDW is associated with inflammatory markers such as C-reactive protein (CRP), erythrocyte sedimentation rate, interleukin-6 and tumor necrosis factor-alpha. Proinflammatory cytokines of sepsis have been shown to suppress the maturation of red blood cells (RBC) and decrease the half-life of RBCs, resulting in the elevation of RDW values Most previous studies investigating the prognostic value of RDW were conducted on adult patients, and similar studies in neonatal sepsis are rare and small. The objective of the present research is to investigate the prognostic role of this routinely available marker in full term neonates with sepsis and to compare it with other traditional prognostic biomarkers.

The prognostic potential of RDW is of particular interest because it is routinely included in the automated complete blood count (CBC) analyses in hospitalized patients and thus available and no additional cost for clinicians.

ELIGIBILITY:
Inclusion Criteria:

* Any infant from birth to 1 month of age with a diagnosis of definite or probable sepsis will included in the study.

Exclusion Criteria:

* gestational age less than 37 weeks.

  * perinatal asphyxia.
  * infants with more than 1 episode of sepsis, only the first one was included.
  * Infants with Dysmorphic features suggestive of chromosomal abnormalities.
  * neonates under a course of antibiotics prior to appropriate blood sampling.

Max Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: - Any infant from birth to 1 month of age with a diagnosis of definite or probable sepsis will included in the study. A diagnosis of definite sepsis is made when a pathogenic agent is isolated from the blood or cerebrospinal fluid in the presence of clinical signs suggestive of sepsis. Probable sepsis is diagnosed when positive cultures are lacking in the presence of signs suggestive of sepsis and 2 positive screening parameters (abnormal CRP, erythrocyte sedimentation rate, platelet count, total leucocytic count, absolute neutrophilic count, or immature/total neutrophils ratio >0.2). When signs of sepsis are existent but both sepsis screening parameters and cultures are negative, this is deemed no sepsis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-02 (Estimated); Primary Completion 2020-01 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
the neonatal mortality rate . | 30 day
  Number of neonates died from sepsis .

CONTACTS AND LOCATIONS:
Overall Officials: Mariam N Gamil, resident, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] Abiodun MT, Oluwafemi RO. Spectrum and outcome of neonatal emergencies seen in a free health-care program in South-Western Nigeria. Niger J Clin Pract. 2017 Mar;20(3):283-289. doi: 10.4103/1119-3077.187324. PMID 28256481
- [Background] Omoigberale AI, Sadoh WE, Nwaneri DU. A 4 year review of neonatal outcome at the University of Benin Teaching Hospital, Benin City. Niger J Clin Pract. 2010 Sep;13(3):321-5. PMID 20857794
- [Background] Tran HT, Doyle LW, Lee KJ, Graham SM. A systematic review of the burden of neonatal mortality and morbidity in the ASEAN Region. WHO South East Asia J Public Health. 2012 Jul-Sep;1(3):239-248. doi: 10.4103/2224-3151.207020. PMID 28615550
- [Background] Liu B, Chen YX, Yin Q, Zhao YZ, Li CS. Diagnostic value and prognostic evaluation of Presepsin for sepsis in an emergency department. Crit Care. 2013 Oct 20;17(5):R244. doi: 10.1186/cc13070. PMID 24138799
- [Background] El Shimi MS, Abou Shady NM, Hamed GM, Shedeed NS. Significance of neutrophilic CD64 as an early marker for detection of neonatal sepsis and prediction of disease outcome. J Matern Fetal Neonatal Med. 2017 Jul;30(14):1709-1714. doi: 10.1080/14767058.2016.1223030. Epub 2016 Aug 31. PMID 27578316
- [Background] Zaki Mel-S, el-Sayed H. Evaluation of microbiologic and hematologic parameters and E-selectin as early predictors for outcome of neonatal sepsis. Arch Pathol Lab Med. 2009 Aug;133(8):1291-6. doi: 10.5858/133.8.1291. PMID 19653728
- [Background] Boskabadi H, Maamouri G, Tavakol Afshari J, Mafinejad S, Hosseini G, Mostafavi-Toroghi H, Saber H, Ghayour-Mobarhan M, Ferns G. Evaluation of serum interleukins-6, 8 and 10 levels as diagnostic markers of neonatal infection and possibility of mortality. Iran J Basic Med Sci. 2013 Dec;16(12):1232-7. PMID 24570828
- [Background] Sadaka F, O'Brien J, Prakash S. Red cell distribution width and outcome in patients with septic shock. J Intensive Care Med. 2013 Sep-Oct;28(5):307-13. doi: 10.1177/0885066612452838. Epub 2012 Jul 17. PMID 22809690
- [Background] Jo YH, Kim K, Lee JH, Kang C, Kim T, Park HM, Kang KW, Kim J, Rhee JE. Red cell distribution width is a prognostic factor in severe sepsis and septic shock. Am J Emerg Med. 2013 Mar;31(3):545-8. doi: 10.1016/j.ajem.2012.10.017. Epub 2013 Feb 4. PMID 23380094
- [Background] Sipahi T, Koksal T, Tavil B, Akar N. The effects of acute infection on hematological parameters. Pediatr Hematol Oncol. 2004 Sep;21(6):513-20. doi: 10.1080/08880010490477301. PMID 15552815
- [Background] Scharte M, Fink MP. Red blood cell physiology in critical illness. Crit Care Med. 2003 Dec;31(12 Suppl):S651-7. doi: 10.1097/01.CCM.0000098036.90796.ED. PMID 14724462
- [Background] Acikgoz SK, Acar B, Aydin S, Acikgoz E, Er O, Sensoy B, Balci MM, Yayla C, Sen F, Topal S, Aydogdu S. Red Cell Distribution Width Can Predict the Significance of Angiographically Intermediate Coronary Lesions. Med Princ Pract. 2016;25(1):31-5. doi: 10.1159/000441001. Epub 2015 Oct 16. PMID 26468646
- [Background] Felker GM, Allen LA, Pocock SJ, Shaw LK, McMurray JJ, Pfeffer MA, Swedberg K, Wang D, Yusuf S, Michelson EL, Granger CB; CHARM Investigators. Red cell distribution width as a novel prognostic marker in heart failure: data from the CHARM Program and the Duke Databank. J Am Coll Cardiol. 2007 Jul 3;50(1):40-7. doi: 10.1016/j.jacc.2007.02.067. Epub 2007 Jun 18. PMID 17601544
- [Background] Li Y, Zhao Y, Feng L, Guo R. Comparison of the prognostic values of inflammation markers in patients with acute pancreatitis: a retrospective cohort study. BMJ Open. 2017 Mar 27;7(3):e013206. doi: 10.1136/bmjopen-2016-013206. PMID 28348184
- [Background] Zhou S, Fang F, Chen H, Zhang W, Chen Y, Shi Y, Zheng Z, Ma Y, Tang L, Feng J, Zhang Y, Sun L, Chen Y, Liang B, Yu K, Jiang S. Prognostic significance of the red blood cell distribution width in diffuse large B-cell lymphoma patients. Oncotarget. 2017 Jun 20;8(25):40724-40731. doi: 10.18632/oncotarget.16560. PMID 28388534
- [Background] Hsieh YP, Tsai SM, Chang CC, Kor CT, Lin CC. Association between red cell distribution width and mortality in patients undergoing continuous ambulatory peritoneal dialysis. Sci Rep. 2017 Apr 3;7:45632. doi: 10.1038/srep45632. PMID 28367961
- [Background] Ramby AL, Goodman DM, Wald EL, Weiss SL. Red Blood Cell Distribution Width as a Pragmatic Marker for Outcome in Pediatric Critical Illness. PLoS One. 2015 Jun 9;10(6):e0129258. doi: 10.1371/journal.pone.0129258. eCollection 2015. PMID 26057629
- [Background] Goldstein B, Giroir B, Randolph A; International Consensus Conference on Pediatric Sepsis. International pediatric sepsis consensus conference: definitions for sepsis and organ dysfunction in pediatrics. Pediatr Crit Care Med. 2005 Jan;6(1):2-8. doi: 10.1097/01.PCC.0000149131.72248.E6. PMID 15636651
- [Background] Minkov GA, Halacheva KS, Yovtchev YP, Gulubova MV. Pathophysiological mechanisms of acute pancreatitis define inflammatory markers of clinical prognosis. Pancreas. 2015 Jul;44(5):713-7. doi: 10.1097/MPA.0000000000000329. PMID 26061557
- [Background] Garofoli F, Ciardelli L, Mazzucchelli I, Borghesi A, Angelini M, Bollani L, Genini E, Manzoni P, Paolillo P, Tinelli C, Merlini G, Stronati M. The red cell distribution width (RDW): value and role in preterm, IUGR (intrauterine growth restricted), full-term infants. Hematology. 2014 Sep;19(6):365-9. doi: 10.1179/1607845413Y.0000000141. Epub 2013 Nov 13. PMID 24225072